CLINICAL TRIAL: NCT01217489
Title: Use of Non-invasive Electrical Impedance Mammography in the Detection, Diagnosis and Characterisation of Breast Lesions
Brief Title: Study Into the Use of Electrical Impedance Mammography in the Diagnosis and Characterisation of Breast Disease
Acronym: Signascan
Status: Terminated | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 09/H0308/12; 07/09/08 V1.3
Record Dates: First submitted 2009-08-18; First posted 2010-10-08 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: breast; cancer; diagnosis; electrical; non-invasive; mammography
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Attendees to symptomatic breast clinic
  Interventions: Procedure: Breast scan - Electrical Impedance Mammography

INTERVENTIONS:
Procedure: Breast scan - Electrical Impedance Mammography — Scanning of the breast on a non-invasive device, using harmless minute electrical currents
  Other Names: Signascan EIM

SUMMARY:
The Signascan Electrical Impedance Mammography (EIM) Study is a pilot study of a non-invasive medical device - a novel approach to breast cancer detection using Electrical Impedance Mammography (passing minute electrical currents through the tissues and detecting the changes to the currents as a result of the tissues, which can differentiate between normal and malignant tissue). The trial is a prospective trial of diagnostic capability of the device, as compared with standard care (diagnosis provided by the concurrent NHS investigation - imaging, surgery etc) performed for female patients attending the symptomatic breast clinic for investigation. The aim is to assess the diagnostic efficacy in detecting 100 true malignancies, and continue to recruit until 300 patients with true malignancies have been recruited if necessary.

DETAILED DESCRIPTION:
Primary Objective

* To test the accuracy of identification of breast malignancy, localisation and tissue characterisation, utilising the non-invasive / non-ionising imaging technique of Electrical Impedance Mammography Secondary Objectives
* Comparative analysis to other imaging modalities for detecting malignant breast disease. Since the Signascan EIM images will be being undertaken in parallel to other imaging modalities it will be possible to perform comparative analyses.
* Determination of whether Electrical Impedance Mammography (EIM) can also be used to identify and tissue-characterise the range of benign clinical breast masses.

Summary of Study Design A pilot study of a system for impedance-based breast screening, designed as a prospective diagnostic pilot study. The procedures for the study will be 'additive', and run in parallel to existing NHS care, therefore no normal investigation or treatment will be withheld. All participant involvement will be during one visit to the hospital, which will be a visit the patient would be making anyway in the course of their routine NHS care pathway. Participation will last only for the time taken to discuss, consent (15 min) and perform (10 min) the scan. Therefore total duration of involvement will be approximately 25 minutes. The pilot study will run for a period of two years, and will aim to include 300 cases of malignant breast disease. Interim analysis will be performed on the first 100 patients. Concepts of blinding/randomization do not apply as they would in a therapeutic trial. Control data will come both from patients' (when normal) contralateral breasts, and from the group of patients scanned but subsequently diagnosed as having benign disease.

5.2 Primary and Secondary Endpoints/Outcome Measures

Primary Outcome Measure:

Determination of success rate of the Signascan EIM method in accurately detecting the presence of malignancy in the breast, and not reporting malignancy in normal breast. (Accuracy' measured as degree of sensitivity (%) and specificity (%) proven in the pilot study population.)

Secondary Outcome Measures:

Determination of ability of the Signascan EIM method to differentiate different types of malignancy (i.e. discerning differences between ductal and lobular carcinoma).

Determination of ability of the Signascan EIM method to differentiate different types of benign tissues (i.e. discerning differences between cystic and fibroadenomatous change).

Study Participants Participants to be included will be women referred for NHS investigation of symptomatic breast lump, following self-examination or picked up by GP. They will generally be in the age range 40-60 years but no eligible patients over 18 yrs will be excluded from the study on the basis of age.

Study Procedures

All study procedures will be performed in one visit scheduled for existing NHS care. Beforehand, where possible, each potential participant will have had a letter and one-page information sheet sent out with the letter inviting them to their NHS appointment. Since 1st January 2010, all referrals to a breast clinic must be seen within 14 days, therefore advance written notice is not possible as many appointments are made by telephone. In these instances patients will be offered a 1 page information sheet when they report to the clinic reception. They will then have time to read and consider it while waiting to be seen and while waiting for investigations to be performed. In these instances judgment will be made by the responsible clinician as to whether it is appropriate to invite the patient to join the study.

In order, the procedures in the clinic (total time 20-25 mins) will be:

1. verbally invite potential participant to study, and go over full-length PIS
2. answer questions and conduct informed consent
3. participant changes into gown
4. position participant on scanning couch
5. push button and perform scan
6. participant dresses and is free to go.

Informed Consent

Written and verbal versions of Informed consent will be presented to the subject detailing no less than: the exact nature of the study; the implications and constraints of the protocol; the known side effects and any risks involved in taking part. It will be clearly stated that the participant is free to withdraw from the study at any time for any reason without prejudice to future care, and with no obligation to give the reason for withdrawal.

The participant will be allowed as much time as wished to consider the information, and the opportunity to question the Principal Investigator, their GP or other independent parties to decide whether they will participate in the study. Written Informed Consent will then be obtained by means of subject dated signature, signature of the person who presented informed consent and, if different, the Principal Investigator (or named Co-Investigator). A copy of the signed Informed Consent will be given to the subject. The original signed form will be retained at the study site.

Study Assessments The assessment confirming eligibility and data necessary for the study will be performed by the participants' ordinary NHS healthcare professionals (the John Radcliffe breast surgery team under Miss Jane Clarke (Consultant breast surgeon) and the associated team of surgeons and nursing staff). The assessment will be as per the standard NHS first-line assessment of symptomatic breast lesions in the population under study. This will tend to include clinical history-taking, clinical breast examination, and standard scanning methods as appropriate. Specific data will be retained for study purposes, including demographic data and other details of medical history and any disease process that may affect the study. This would include breast disease in either breast, prior surgery, and significant systemic comorbidities. Additionally, since hormone status may affect the impedance profiles of breast tissue, data on dates of menstrual cycles will be collected also. Miss Clarke and team will identify and approach suitable patients to invite them to join the study, on their assessment visit.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Female, aged 18 years or above
* Attending for investigation of symptomatic breast lump

Exclusion Criteria:

* Pacemaker or critical implanted electronic device
* Under the age of 18 years
* Adults with learning disabilities
* Adults who are unconscious or very severely ill
* Adults who have a terminal illness
* Adults in emergency situations
* Adults suffering from a mental illness
* Adults with dementia
* Prisoners
* Young offenders
* Adults who are unable to consent for themselves
* Any person considered to have a particularly dependent relationship with investigators
* Any others deemed to belong to a vulnerable group

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants to be included will be women referred for NHS investigation of symptomatic breast lump, following self-examination or picked up by GP. They will generally be in the age range 40-60 years but no eligible patients over 18 yrs will be excluded from the study on the basis of age.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-03-01 (Actual); Study Completion 2012-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Clarke, Mb BCh, Principal Investigator — Oxford Radcliffe Hospitals NHS Foundation Trust
Locations (1):
- Oxford Radcliffe Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom